CLINICAL TRIAL: NCT03157154
Title: Bleeding Risk Evaluation in Haemophilia Patients Under Antiplatelet Therapies
Acronym: ERHEA
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC17_0150
Record Dates: First submitted 2017-05-16; First posted 2017-05-17 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Hemophilia
Keywords: Haemophilia; Atherosclerosis; Atrial fibrillation; Antiplatelets; Anticoagulant
MeSH Terms: conditions — Hemophilia A; Atherosclerosis; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- First group: Haemophilia patients with history of either cardiovascular disease or atrial fibrillation undergoing an antiplatelet or anticoagulant prophylaxis
  Interventions: Other: Non interventional study
- Control group: Haemophilia patient without such history or treatment matched on age and disease status (haemophilia A or B and the severity of the disease : severe, mild, minor).
  Interventions: Other: Non interventional study

INTERVENTIONS:
Other: Non interventional study — A query form to all concerned patients by each investigating centre will be send

SUMMARY:
Life expectancy of haemophilia patients (specially severe) has dramatically increase in the last decades, which lead to the apparition of aging diseases such as cardiovascular disease, with the potential bleeding risk of antiplatelet therapies and anticoagulants.

The primary endpoint of the study is to evaluate this bleeding risk in haemophilia patients (all severity) with such treatment in comparison to non treated patients, according to the number of bleeding events in the last year reported by the haemophilia patients under study treatment (antiplatelet and anticoagulant) in comparison to haemophilia patients free of such treatment. The main hypothesis is that antiplatelet and anticoagulant therapy can be safely used in minor haemophilia patients but might lead to increase bleeding risk in other haemophilia patients.

Secondary endpoint consist in:

* Evaluate the impact of know cardio-vascular risk in haemophilia patients (Odd ratios=OR)
* Evaluate the number of sever bleeding event in patient under study treatments compared to the control group
* Evaluate the overall consumption of factor VIII or IX supply in patients under study treatments compared to control group
* Estimate the stenosis relapse risk in haemophilia patients with arterial STENT
* Estimate the embolic risk of haemophilia patients with atrial fibrillation

Population description:

Haemophilia patients (man, all severity)

Age above 50 years, followed during the last 5 years in one of the study centre

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age above 50 years
* Hemophilia A or B carriers
* Followed within the 5 last years in one of the research center

Exclusion Criteria:

* Jurisdictional prevention procedures
* Other medical condition that might interfere with the bleeding risk (Willebrand's disease, Other coagulation factor deficiencies, haematological malignancies, …)
* Other drugs that might interfere with the bleeding risk (Serotonin reuptake inhibitors)
* Patient refusal

Min Age: 50 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Haemophilia patients (man, all severity)
  Age above 50 years, followed during the last 5 years in one of the study centre
Sampling Method: Non-Probability Sample
Enrollment: 259 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
Number of bleeding occurrences | last 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Marc Trossaërt, Dr, Principal Investigator — Nantes University Hospital
Locations (6):
- France (6):
  - Angers University Hospital, Angers
  - Brest University Hospital, Brest
  - Le Mans Hospital, La Mans
  - Lyon University Hospital, Lyon
  - Rennes University Hospital, Rennes
  - Tours University Hospital, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Desjonqueres A, Guillet B, Beurrier P, Pan-Petesch B, Ardillon L, Pineau-Vincent F, Sigaud M, Fouassier M, Ternisien C, Gillet B, Bene MC, Horvais V, Lienhart A, Trossaert M. Bleeding risk for patients with haemophilia under antithrombotic therapy. Results of the French multicentric study ERHEA. Br J Haematol. 2019 May;185(4):764-767. doi: 10.1111/bjh.15606. Epub 2018 Oct 18. No abstract available. PMID 30338508